CLINICAL TRIAL: NCT07241559
Title: Comparison of the Effectiveness of Thoracolumbar Fascia Mobilization and Ultrasound-Guided Thoracolumbar Interfascial 5% Dextrose Injection in Patients With Chronic Low Back Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Collaborators: Ankara Training and Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025/5
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Chronic Low Back Pain
Keywords: Dextrose Injection; Mobilization; Thoracolumbar Fascia
MeSH Terms: interventions — Glucose; Myofascial Release Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Thoracolumbar Fascia Mobilization Group (Active Comparator): Patients in this group will receive thoracolumbar fascia mobilization. A total of six sessions of myofascial release therapy will be administered twice per week for three weeks.
  Interventions: Procedure: Myofascial Release
- Thoracolumbar Interfascial 5% Dextrose Injection Group (Active Comparator): Patients in this group will receive ultrasound-guided thoracolumbar interfascial 5% dextrose injection.
  After being informed about the procedure, the patient will be placed in the prone position on the examination table, with a small pillow placed under the abdomen to allow relaxation of the lumbar muscles.
  Axial scanning will be performed using a Logiq 9 (GE Medical Systems®) ultrasound device equipped with a linear probe (7-12 MHz, "ZONARE"), and the probe will be positioned at the level of the L3 spinous process. The multifidus, longissimus, and iliocostalis muscles will be visualized.
  A 21-gauge (0.80 × 38 mm) needle will then be inserted from lateral to medial into the interfascial plane of the posterior layer of the thoracolumbar fascia using an in-plane technique. After confirming negative aspiration (to rule out vascular puncture), 10 mL of 5% dextrose solution will be injected into the target area.
  Interventions: Drug: 5% Dextrose
- Combined Therapy Group (Active Comparator): Patients in this group will receive both myofascial release therapy and ultrasound-guided thoracolumbar interfascial 5% dextrose injection as described above.
  Interventions: Drug: 5% Dextrose; Procedure: Myofascial Release

INTERVENTIONS:
Drug: 5% Dextrose — 10 mL of 5% dextrose solution will be injected into the target area.
  Arms: Combined Therapy Group; Thoracolumbar Interfascial 5% Dextrose Injection Group
Procedure: Myofascial Release — Patients in this group will receive thoracolumbar fascia mobilization. A total of six sessions of myofascial release therapy will be administered twice per week for three weeks.
  Arms: Combined Therapy Group; Thoracolumbar Fascia Mobilization Group

SUMMARY:
The aim of this study is to investigate the effects of thoracolumbar fascia mobilization and ultrasound-guided thoracolumbar interfascial 5% dextrose injection on pain, range of motion, disability, quality of life, proprioception, and fascial thickness and echogenicity in patients with nonspecific chronic low back pain.

-Primary Objective: The primary objective is to evaluate the effects of these interventions on pain, functional status and range of motion.

-Secondary Objective: The secondary objective is to assess the long-term effects on quality of life, proprioception, fascial thickness, and echogenicity.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged 18 to 65 years
2. Presence of low back pain lasting longer than 3 months
3. No adequate response to medical treatment
4. Voluntary participation in the study

Exclusion Criteria:

1. Age below 18 or above 65 years
2. Body mass index (BMI) greater than 30 kg/m²
3. Pregnancy or breastfeeding
4. Presence of coagulation disorders
5. History of spinal surgery
6. Presence of inflammatory or malignant diseases
7. Local infection at the spine or injection site
8. Presence of lumbar disc pathology causing radiculopathy
9. Presence of spinal stenosis, spondylolysis, or spondylolisthesis
10. Participation in physical therapy or any manual therapy within the past 6 months
11. Receiving lumbar injections within the past 6 months
12. History of allergy to injection materials
13. Refusal to participate in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-05-20 (Actual); Primary Completion 2025-11-20 (Estimated); Study Completion 2026-02-20 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | Baseline, after 1 month and 3 month changes
  Patients' back pain scores will be recorded using a VAS (Visual Analog Scale). The VAS method used to assess pain intensity is a scale from 0 (no pain) to 10 (unbearable pain), with the patient selecting the number that corresponds to their pain.
Lumbar spine range of motion (ROM) | Baseline, after 1 month and 3 month changes
  Lumbar spine range of motion (ROM) was evaluated using both a dual digital inclinometer and the Modified Schober Test.
  For the inclinometer assessment, a dual digital inclinometer (Baseline® Digital Inclinometer, Fabrication Enterprises Inc., USA) was used. Participants were positioned in a standing posture with feet shoulder-width apart and knees fully extended. The spinous processes of T12 and S1 vertebrae were palpated and marked as anatomical reference points.
  Two inclinometers were placed over these landmarks-one at T12 and one at S1-and both were zeroed in the neutral position. Participants were instructed to perform lumbar flexion, extension, and lateral flexion slowly without bending the knees or rotating the pelvis.
  The lumbar ROM for each direction was calculated as the difference between the angular readings at T12 and S1 levels. Each movement was measured three times, and the mean value was used for analysis.
  Additionally, lumbar flexion was also assessed using the Modif
Functional Status Assessment (Oswestry Disability Index - ODI) | Baseline, after 1 month and 3 month changes
  Functional status was assessed using the Oswestry Disability Index (ODI), one of the most commonly used and validated questionnaires for evaluating disability related to low back pain.
  The ODI consists of 10 sections, each addressing a different aspect of daily living affected by back pain, including pain intensity, personal care, lifting, walking, sitting, standing, sleeping, social life, traveling, and employment or homemaking.
  Each item is scored on a 6-point Likert scale ranging from 0 (no disability) to 5 (maximum disability).
  The total score is calculated by summing the responses, dividing by the maximum possible score, and multiplying by 100 to obtain a percentage of disability.
  Higher scores indicate greater functional limitation.
  Participants completed the ODI questionnaire at baseline and after the intervention to assess changes in functional status over time.

SECONDARY OUTCOMES:
Quality of Life Assessment (SF-12 Health Survey) | Baseline, after 1 month and 3 month changes
  Quality of life was assessed using the 12-Item Short Form Health Survey (SF-12), a validated and widely used self-reported questionnaire designed to evaluate overall health status.
  The SF-12 measures both physical and mental health components, summarized as the Physical Component Summary (PCS) and Mental Component Summary (MCS) scores.
  Participants completed the SF-12 questionnaire at baseline and after the intervention. Each item was scored according to the standardized SF-12 scoring algorithm, and results were converted into normalized scores (mean = 50, SD = 10) to allow comparison with general population norms.
  Higher scores indicate better perceived health status and quality of life. The SF-12 has been validated for use in musculoskeletal and chronic pain populations and is suitable for evaluating treatment-related changes in functional health and well-being.
Thoracolumbar Fascia Thickness and Echogenicity Assessment | Baseline, after 1 month and 3 month changes
  Thoracolumbar fascia (TLF) morphology was evaluated using ultrasound imaging, following the methodology described by Langevin et al. The ultrasound probe was positioned transversely at the L2-L3 interspinous level, where the thoracolumbar fascia lies parallel to the skin surface.
  High-resolution B-mode ultrasound images of the thoracolumbar fascia were obtained and recorded for each participant under standardized conditions.
  The thickness and echogenicity of the fascia were analyzed using ImageJ® software (National Institutes of Health, USA), a freely available image processing program.
  Fascial thickness was measured as the distance between the superficial and deep fascial borders, and echogenicity was quantified using grayscale intensity analysis within a standardized region of interest (ROI).
  All ultrasound assessments were performed by the same experienced physiatrist to ensure measurement reliability.
Lumbar Proprioception Assessment | Baseline, after 1 month and 3 month changes
  Lumbar proprioception was evaluated using an active joint position sense test performed in the sitting position.
  Participants were seated comfortably with their pelvis stabilized and were instructed to move their trunk from a neutral starting position to a predetermined target angle in the sagittal plane (flexion or extension).
  After reaching the target position, participants maintained the posture for a few seconds to familiarize themselves with it, then returned to the starting (neutral) position.
  Following three practice trials involving maximal flexion and extension, each participant was asked to reproduce the target position without visual feedback.
  The repositioning error-the difference between the target angle and the angle reproduced by the participant-was measured using a universal goniometer.
  Three measurements were obtained, and the mean repositioning error was recorded for analysis.
  Smaller errors indicated better proprioceptive accuracy.

CONTACTS AND LOCATIONS:
Overall Officials: Büşra ALÇIN, Medical Doctor, Principal Investigator — Ankara Training and Research Hospital; Nida KOÇER NAZLIGÜL, Medical Doctor, Study Director — Ankara Training and Research Hospital; Barış NACIR, Study Director — Ankara Training and Research Hospital
Locations (1):
- Ankara Training and Research Hospital, Ankara, Altındağ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Langevin HM, Fox JR, Koptiuch C, Badger GJ, Greenan-Naumann AC, Bouffard NA, Konofagou EE, Lee WN, Triano JJ, Henry SM. Reduced thoracolumbar fascia shear strain in human chronic low back pain. BMC Musculoskelet Disord. 2011 Sep 19;12:203. doi: 10.1186/1471-2474-12-203. PMID 21929806